CLINICAL TRIAL: NCT04532996
Title: Trauma-focused Psychodynamic Psychotherapy for LGBT Patients With Post-traumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-05022019
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-10

CONDITIONS: Complex Post-Traumatic Stress Disorder; Post-traumatic Stress Disorder
Keywords: PTSD; psychotherapy; psychodynamic; LGBTQ
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — 2,2,3,3-tetrafluoroputrescine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trauma-focused psychodynamic psychotherapy (Experimental): Twice-weekly psychotherapy for 20-24 sessions.
  Interventions: Behavioral: Trauma-focused psychodynamic psychotherapy

INTERVENTIONS:
Behavioral: Trauma-focused psychodynamic psychotherapy — This psychotherapy addresses disruptions in narrative coherence and affective dysregulation by exploring the psychological meanings of symptoms and their relation to traumatic events. The therapist works to identify intrapsychic conflicts, intense negative affects, and defense mechanisms related to the PTSD syndrome using a psychodynamic formulation that provides a framework for intervention. The transference provides a forum for patients to address feelings of mistrust, difficulties with authority, fears of abuse, angry and guilty feelings, and fantasies.
  This treatment will be provided in-person or over teletherapy as the public health situation demands.
  Other Names: TFPP

SUMMARY:
This is a pilot, open trial of trauma-focused psychodynamic psychotherapy for LGBT-identifying individuals who meet for DSM-5 defined post-traumatic stress disorder and are interested in receiving a research psychotherapy intervention. A sample of at least 15 therapy completers will be collected.

DETAILED DESCRIPTION:
Despite high prevalence of PTSD among LGBT individuals, there are no data characterizing the disorder in this population, nor its treatment. This represents an important under-researched area in LGBT care and treatment. The purpose of this study is: (a) to preliminarily characterize PTSD within an LGBT sample; and (b) to test out the preliminary effects and acceptability of a novel PTSD psychotherapy, trauma-focused psychodynamic psychotherapy, in this group. Participants identifying as LGBT and meeting DSM-5 criteria for PTSD per a structured, reliable clinical interview for PTSD will receive 20-24 sessions of twice-weekly TFPP at no cost. Participants will receive four detailed clinical research assessments, at baseline/study entry, Week 5 of treatment, treatment termination/end (Week 12), and 3-months after the end of treatment.

TFPP is adapted from the only empirically supported, non-exposure focused psychodynamic therapy for panic disorder and anxiety disorders, panic-focused psychodynamic psychotherapy. TFPP aims to improve patients' ability to understand and manage strong, intense emotions that appear seemingly "out of the blue," which links to their tendency to reexperience traumatic events in the here-and-now. TFPP addresses the psychological meanings of symptoms and their relationship to traumatic events to help the patient understand underlying emotions triggering their symptoms and the ways in which trauma influences their current experiences. TFPP was developed for patients with complex PTSD, who often have multiple prior trauma exposures with no clear "index" trauma. Moreover, TFPP also explicitly considers opportunities for patients to explore the broader context of their symptoms and difficulties, including but not limited to LGBT identity or experiences of oppression.

ELIGIBILITY:
Inclusion Criteria:

* Identify as LGBTQ
* CAPS-5 diagnosed PTSD per DSM-5 criteria
* Stable medication for >=2 months and ongoing during treatment

Exclusion Criteria:

* Psychosis or bipolar disorder
* Primary substance use disorder
* Severe suicidality
* Severe depression per a reconstructed Hamilton Rating Scale for Depression score of >=24
* Organic mental syndromes interfering with trial demands

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Treatment Response on Clinician Administered PTSD Scale for DSM-5 | Baseline (to calculate what is defined as a 30% change from initial CAPS severity score), Mid-Treatment (Week 5), Termination (Week 12), Follow-Up (3 Months Post Treatment)
  The CAPS is the gold-standard measure for PTSD symptoms and diagnosis given by trained research assistants; lower scores denote less severe PTSD symptoms; a decline of at least 30% from an individual's baseline CAPS score is defined as a treatment response on the CAPS.

SECONDARY OUTCOMES:
Attrition from treatment by end of therapy duration (Week 12) | Anytime between Baseline and Termination (Week 12)
  Failure to complete experimental psychotherapy intervention (defined as attending at least 16 out of 24 TFPP sessions within the 12-week period OR patient declaring intention to not attend any further TFPP sessions during the 12-week period). The specific session in which the patient dropped out will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: John R Keefe, PhD, Principal Investigator — Weill Medical College of Cornell University / NYP-Weill Cornell
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Milrod B, Keefe JR, Choo TH, Arnon S, Such S, Lowell A, Neria Y, Markowitz JC. Separation anxiety in PTSD: A pilot study of mechanisms in patients undergoing IPT. Depress Anxiety. 2020 Apr;37(4):386-395. doi: 10.1002/da.23003. Epub 2020 Feb 25. PMID 32097526
- [Background] Busch FN, Nehrig N, Milrod B. Trauma-Focused Psychodynamic Psychotherapy of a Patient With PTSD in a Veterans Affairs Setting. Am J Psychother. 2019 Mar 1;72(1):24-28. doi: 10.1176/appi.psychotherapy.20180019. Epub 2019 Feb 21. PMID 30786735
- [Background] Busch FN, Milrod BL. Trauma-Focused Psychodynamic Psychotherapy. Psychiatr Clin North Am. 2018 Jun;41(2):277-287. doi: 10.1016/j.psc.2018.01.005. PMID 29739526